CLINICAL TRIAL: NCT07046988
Title: Population Pharmacokinetics of Terbinafine in Children With Tinea Capitis
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: SDU-ZW-PPK-014
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Tinea Capitis
Keywords: Tinea Capitis
MeSH Terms: conditions — Tinea Capitis | interventions — Terbinafine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Terbinafine Tablets — Oral administration once daily:
  For patients weighing <20 kg: 62.5 mg qd; For patients weighing 20-40 kg: 125 mg qd; For patients weighing >40 kg: 250 mg qd; Total 8 weeks.

SUMMARY:
The goal of this observational study is to characterize the population pharmacokinetics (PPK) of terbinafine in pediatric patients with tinea capitis, evaluate its efficacy and safety, and identify covariates affecting drug disposition in Chinese children aged 2-18 years diagnosed with tinea capitis and treated with oral terbinafine. The main questions it aims to answer are:

What are the terbinafine pharmacokinetic parameters (e.g., AUC, CL, V) in children with tinea capitis, and how do they differ from adult values? Which covariates (e.g., age, body weight, CYP enzyme activity, renal function) significantly influence inter-individual variability in terbinafine PK parameters? What is the clinical efficacy (based on TSSS reduction and mycological cure rate) and safety profile of terbinafine in this pediatric population?

Participants will:

Undergo oral terbinafine treatment according to weight-based dosing (62.5-250 mg daily).

Concentration determination is carried out using the opportunistic sampling method.

Complete clinical assessments (TSSS scoring) and mycological examinations (microscopy/culture) at baseline and follow-up visits.

Undergo routine laboratory tests (liver/kidney function, hematology) to monitor safety.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 2 to 18 years;
2. Diagnosis of tinea capitis:

   * Typical clinical manifestations, dermatoscopic findings combined with Wood's lamp examination; ② Positive mycological examination, including positive fungal microscopy and/or isolation of dermatophytes by fungal culture; ③ Exclusion of scalp seborrheic dermatitis, psoriasis, alopecia areata, lupus erythematosus, lichen planopilaris, trichotillomania, suppurative perifolliculitis of scalp, syphilitic alopecia, etc.

Exclusion Criteria:

1. Concomitant topical treatment with terbinafine;
2. Conditions interfering with gastrointestinal absorption of terbinafine;
3. Documented hepatic/renal impairment or hematological disorders;
4. Receipt of radiotherapy, systemic cytostatic/immunosuppressive therapy, or antibacterial/antiviral/antiparasitic therapy currently or within 2 weeks prior to study initiation;
5. Participation in other clinical trials, or other circumstances deemed inappropriate by the investigator.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Chinese pediatric patients aged 2 to 18 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Terbinafine concentration | Through study completion, an average of 12 weeks.
  Terbinafine plasma concentration, terbinafine concentration in hair
AUC | Through study completion, an average of 12 weeks.
  Area under the curve (AUC)
CL | Through study completion, an average of 12 weeks.
  Clearance (CL)
V | Through study completion, an average of 12 weeks.
  Apparent volume of distribution (V)
CV% | Through study completion, an average of 12 weeks.
  Inter-individual variability (CV%) of AUC, CL and V with covariates

SECONDARY OUTCOMES:
Clinical Efficacy | The end of fellow-up, at 12 weeks
  Defined as a 60-99% reduction in TSSS compared to baseline. Values below 60% are considered ineffective.
  Clinical efficacy rate = (number of effective cases / total cases) × 100%. TSSS is a scale scoring the severity of 5 signs and symptoms (erythema, desquamation/scaling, papules, pustules, and pruritus) into 4 grades (0 = none; 1 = mild; 2 = moderate; 3 = severe). The sum of these scores yields TSSS, with a maximum of 15 points.
Clinical Cure | The end of fellow-up, at 12 weeks
  Defined as 100% efficacy (TSSS = 0). Clinical cure rate = (number of clinically cured cases / total cases) × 100%. TSSS is a scale scoring the severity of 5 signs and symptoms (erythema, desquamation/scaling, papules, pustules, and pruritus) into 4 grades (0 = none; 1 = mild; 2 = moderate; 3 = severe). The sum of these scores yields TSSS, with a maximum of 15 points.
Mycological Cure | The end of fellow-up, at 12 weeks
  Defined as negative mycological examination results. Mycological cure rate = (number of mycologically cured cases / total cases) × 100%.
Safety Assessment Indicators | From enrollment to the end of treatment about 12 weeks
  Drug-related adverse events and serious adverse events during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided